CLINICAL TRIAL: NCT00001114
Title: A Randomized Phase II Trial to Determine the Safety, Tolerance, and Efficacy of Two Doses of Interferon Alfa-2b Combined With Didanosine in Patients With Kaposi's Sarcoma
Brief Title: The Safety and Effectiveness of Interferon Alfa-2B Plus Didanosine in Patients With Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Schering-Plough (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 206; 11183 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Didanosine; Drug Interactions; Acquired Immunodeficiency Syndrome; Interferon-alpha
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Interferon alpha-2; Didanosine

INTERVENTIONS:
Drug: Interferon alfa-2b
Drug: Didanosine

SUMMARY:
Primary: To evaluate the safety, toxicity, and antitumor activity of two doses of interferon alfa-2b (IFN-alpha) combined with a fixed dose of didanosine (ddI) in patients with Kaposi's sarcoma associated with HIV infection.

Secondary: To evaluate the effects of combined IFN-alpha and ddI treatment on HIV expression and markers of immune function.

Previous studies have shown that IFN-alpha can induce regression of Kaposi's sarcoma and suppression of HIV in some patients. Although various trials using IFN-alpha in combination with the nucleoside analogue zidovudine have demonstrated a high degree of antitumor activity and evidence of HIV suppression, the overlapping toxicity (primarily neutropenia) of these two agents has proven dose-limiting. The toxicity profile of ddI suggests that this drug may be better tolerated than zidovudine when combined with IFN-alpha.

DETAILED DESCRIPTION:
Previous studies have shown that IFN-alpha can induce regression of Kaposi's sarcoma and suppression of HIV in some patients. Although various trials using IFN-alpha in combination with the nucleoside analogue zidovudine have demonstrated a high degree of antitumor activity and evidence of HIV suppression, the overlapping toxicity (primarily neutropenia) of these two agents has proven dose-limiting. The toxicity profile of ddI suggests that this drug may be better tolerated than zidovudine when combined with IFN-alpha.

Up to 90 patients are randomized to receive either low or high doses of IFN-alpha (1 or 10 million Units/day) in combination with a fixed dose of ddI. Fourteen patients are initially entered at each dose level. If no objective antitumor responses are observed among the first 14 patients at a given dose, no further patients are entered on that treatment arm. If one or more antitumor responses are seen at a given dose, up to 45 patients may be entered on that treatment arm. Patients must complete at least 4 weeks of study therapy to be considered evaluable for tumor response. Treatment is continued until tumor progression or unacceptable toxicity occurs. PER AMENDMENT 9/19/96: NOTE - After 16 weeks of treatment subjects may receive any FDA approved antiretroviral drug regimen in addition to or in place of ddI.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Chemoprophylaxis for candidiasis and herpes simplex.
* Up to 14 days of metronidazole.
* Recombinant erythropoietin.
* G-CSF (for severe cases of neutropenia).
* Isoniazid for treatment of TB if given in conjunction with pyridoxine.

Required in patients with CD4 counts < 200 cells/mm3:

* Prophylaxis for PCP.

PER AMENDMENT 9/19/96:

* After the first 16 weeks of combined IFN alpha-2b and ddI treatment subjects may at the discretion of the investigator receive any FDA approved antiretroviral drug regimen in addition to or in place of ddI.

Patients must have:

* Positive antibody to HIV.
* Biopsy-proven Kaposi's sarcoma (at least 5 measurable lesions, with at least 1 measurable cutaneous lesion) involving the skin, lymph nodes, oral cavity, or asymptomatic lesions of the GI tract not requiring systemic chemotherapy. Lung involvement with Kaposi's sarcoma excludes.
* Consent of parent or guardian if less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Concurrent opportunistic infection or B symptoms including unexplained fever, night sweats, weight loss > 10 percent, and diarrhea lasting more than 2 weeks.
* Visceral (non-nodal) Kaposi's sarcoma requiring cytotoxic chemotherapy.
* Severe (> 2+) tumor-associated edema.
* Concurrent neoplasia other than basal cell carcinoma, or anogenital intraepithelial neoplasia.
* Current clinical evidence of peripheral neuropathy (= or > grade 1), pancreatitis, intractable diarrhea, or active seizure disorder not well controlled by anti-seizure medications.
* Significant symptomatic cardiac disease.
* Medical contraindication.

Concurrent Medication:

Excluded:

* Other investigational, antiviral, immunomodulating, or antitumor agents.
* Drugs associated with peripheral neuropathy (other than ddI).

PER AMENDMENT 9/19/96:

* Other antiretroviral agents may not be taken during the first 16 weeks of combined IFN alpha-2b and ddI treatment.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following prior conditions are excluded:

* Opportunistic infection or B symptoms including unexplained fever, night sweats, weight loss > 10 percent, and diarrhea lasting more than 2 weeks.
* Prior grade 3 or 4 toxicity attributed to ddI therapy.
* Prior history of peripheral neuropathy (= or > grade 1), pancreatitis, intractable diarrhea, or active seizure disorder not well controlled by anti-seizure medications.
* History of myocardial infarction or ventricular arrhythmias.

Prior Medication:

Excluded:

* Prior IFN-alpha.
* Corticosteroids, biological response modifiers, cytotoxic chemotherapy, or known neurotoxic drugs (other than ddI or ddC) within 30 days prior to study entry.
* Therapy with antiretroviral drugs (other than ddI) within 7 days prior to study entry.

Prior Treatment:

Excluded:

* Radiation therapy within 30 days prior to study entry.

Risk Behavior:

* Alcohol consumption is strongly discouraged.
* Patients considered to be noncompliant should be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krown SE, Study Chair
Locations (13):
- United States (12):
  - Stanford CRS, Palo Alto, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Bmc Actg Crs, Boston, Massachusetts
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Krown SE, Li P, Von Roenn JH, Paredes J, Huang J, Testa MA. Efficacy of low-dose interferon with antiretroviral therapy in Kaposi's sarcoma: a randomized phase II AIDS clinical trials group study. J Interferon Cytokine Res. 2002 Mar;22(3):295-303. doi: 10.1089/107999002753675712. PMID 12034036